CLINICAL TRIAL: NCT01443689
Title: A Phase Ι/Π Study of Human Cord Blood Mononuclear Cells and Human Umbilical Cord Mesenchymal Stem Cells Transplantation in Patients With Acute Burn
Brief Title: Allogenic Stem Cell Therapy in Patients With Acute Burn
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BKCR-BURN-1.0(2011)
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Burns
Keywords: Extensive Burn; Human Cord Blood Mononuclear Cells; Human Umbilical Cord Mesenchymal Stem Cells
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group1 :Conventional plus hUCMSCs treatment (Experimental): Participants will be given conventional therapy plus human cord mesenchymal stem cells transplantation with a 6 months follow-up.
  Interventions: Biological: human umbilical cord mesenchymal stem cells
- Group 2: Conventional plus hCBMNCs and hUCMSCs therapy (Experimental): Participants will be given conventional therapy plus combination of hCBMNCs together with hUCMSCs transplantation with a 6 months follow-up.
  Interventions: Biological: human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells
- Group 3:Conventional therapy (Active Comparator): Participants will be given conventional therapy only with a 6 months follow-up.
  Interventions: Drug: Conventional therapy

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells — Participants will be given conventional therapy plus hUCMSCs transplantation.
  Arms: Group1 :Conventional plus hUCMSCs treatment
Biological: human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells — Participants will be given conventional therapy plus and hCBMNCs and hUCMSCs transplantation.
  Arms: Group 2: Conventional plus hCBMNCs and hUCMSCs therapy
Drug: Conventional therapy — Participants will be given conventional therapy only.
  Arms: Group 3:Conventional therapy

SUMMARY:
Burn trauma,especially extensive ones, remains a life-threatening local and general inflammatory condition destroying the skin and underlying tissues, and resulting in serious sequelae. Remarkable progress has been achieved during last 30 years，stem cell therapy plays an important role in this progress. Human umbilical cord mesenchymal stem cells (hUCMSCs) and human cord blood mononuclear cells (hCBMNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy for burn. In this study, the safety and efficacy of hUCMSCs and hCBMNCs transplantation will be evaluated in patients with acute burn.

DETAILED DESCRIPTION:
To investigate the safety and efficacy of human cord blood mononuclear cells and human umbilical cord mesenchymal stem cells transplantation in patients of Acute, Moderate-Severe, Full-thickness burn.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18- 65 years, both gender.
* Diagnosed with Acute, Moderate-Severe, full-thickness burn:

Burn occurring within the 72 hours prior to administration. TBSA 20-55%, third degree wounds surface area < 19 % ;

* Willing to sign the Informed Consent Form.

Exclusion Criteria:

* All other burns except thermal origin.
* Chronically malnourished, poor medical condition or shock
* Systemic inflammatory response syndrome (SIRS) or septicopyemia
* Moderate-severe inhalation injury airways to lung
* HIV+
* Autoimmune disease, e.g. lupus erythematosus, multiple sclerosis.
* Severe pulmonary and hematological disease, malignancy or hypo-immunity.
* Currently undertaking other treatment that may affect the safety/efficacy of stem cells.
* Pregnancy or lactation
* Enrollment in other trials in the last 3 months.
* Other criteria the investigator consider improper for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The ratio of wound contraction and re-epithelialisation | 6 months after treatment
Complete healing time for investigated burn area | 6 months after treatment
Vancouver Scar Scale | 6 months after treatment

SECONDARY OUTCOMES:
Incidence of infections and bleedings in burn wounds | 6 months after treatment]
Engraftment assessment: Vitality of the graft | 6 months after treatment]
McGill pain Questionnaire | 6 months after treatment
Incidence of Adverse Events and Serious Adverse Events | 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Kunmming Medical College, Kunming, Yunnan, China